CLINICAL TRIAL: NCT02406781
Title: Combination of MK3475 and Metronomic Cyclophosphamide in Patients With Advanced Sarcomas : Multicentre Phase II Trial
Acronym: PEMBROSARC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Ministry of Health, France (Other Government); Immune Design, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB 2014-04; 2014-004568-39 (EudraCT Number)
Record Dates: First submitted 2015-03-12; First posted 2015-04-02 (Estimated); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Sarcoma
Keywords: Efficacy of MK 3475 with Metronomic Cyclophosphamide; Advanced Sarcomas; Leiomyosarcoma; Undifferentiated Sarcoma; Other Sarcoma; GIST; Osteosarcoma
MeSH Terms: conditions — Sarcoma; Leiomyosarcoma; Osteosarcoma | interventions — pembrolizumab; Cyclophosphamide; TLR4 agonist G100

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Stratum 1: Advanced Leiomyosarcoma (Experimental): Treatment strategy A: Combination of MK3475 with Metronomic CP administered to patients with advanced leiomyosarcoma.
  MK3475 will be administered intraveinously. Metronomic CP (Cyclophosphamide) will be adminstered orally.
  Interventions: Drug: Combination of MK3475 with Metronomic CP
- Stratum 2: Advanced undifferentiated sarcoma (Experimental): Treatment strategy A: Combination of MK3475 with Metronomic CP administered to patients with advanced undifferentiated sarcoma.
  MK3475 will be administered intraveinously. Metronomic CP (Cyclophosphamide) will be adminstered orally.
  Interventions: Drug: Combination of MK3475 with Metronomic CP
- Stratum 3: Advanced other sarcoma (Experimental): Treatment strategy A: Combination of MK3475 with Metronomic CP administered to patients with advanced other sarcoma.
  MK3475 will be administered intraveinously. Metronomic CP (Cyclophosphamide) will be adminstered orally.
  Interventions: Drug: Combination of MK3475 with Metronomic CP
- Stratum 4: Advanced osteosarcoma (Experimental): Treatment strategy A: Combination of MK3475 with Metronomic CP administered to patients with advanced osteosarcoma.
  MK3475 will be administered intraveinously. Metronomic CP (Cyclophosphamide) will be adminstered orally.
  Interventions: Drug: Combination of MK3475 with Metronomic CP
- Stratum 5: Advanced GIST (Experimental): Treatment strategy A: Combination of MK3475 with Metronomic CP administered to patients with advanced GIST.
  MK3475 will be administered intraveinously. Metronomic CP (Cyclophosphamide) will be adminstered orally.
  Interventions: Drug: Combination of MK3475 with Metronomic CP
- Stratum 6: Advanced soft-tissue sarcomas with immune signature (Experimental): Treatment strategy A: Combination of MK3475 with Metronomic CP administered to patients with advanced soft-tissue sarcomas with immune signature.
  MK3475 will be administered intraveinously. Metronomic CP (Cyclophosphamide) will be adminstered orally.
  Interventions: Drug: Combination of MK3475 with Metronomic CP
- Stratum 7: Metastatic soft-tissue sarcoma. (Experimental): Treatment strategy B: Combination of MK3475 with Metronomic CP and G100 adminitrered to patients with metastatic soft-tissue sarcoma.
  MK3475 will be administered intravenously. Metronomic CP (Cyclophosphamide) will be administered orally. G100 will be administered by intra-tumoral injection.
  Interventions: Drug: Combination of MK3475 with Metronomic CP and G100

INTERVENTIONS:
Drug: Combination of MK3475 with Metronomic CP — Combination of MK3475 with Metronomic CP. Metronomic CP (cyclophosphamide) will be administered per os bi-daily (50 mg x 2), and given on a week on/ week off schedule.
  MK3475 will be administered intraveinously, and given every 3 weeks on day 8. A treatment cycle consists of 3 weeks. Treatment may continue until disease progression or study discontinuation.
  Other Names: Pembrolizumab, Endoxan
  Arms: Stratum 1: Advanced Leiomyosarcoma; Stratum 2: Advanced undifferentiated sarcoma; Stratum 3: Advanced other sarcoma; Stratum 4: Advanced osteosarcoma; Stratum 5: Advanced GIST; Stratum 6: Advanced soft-tissue sarcomas with immune signature
Drug: Combination of MK3475 with Metronomic CP and G100 — Combination of MK3475 with Metronomic CP and G100. Metronomic CP (cyclophosphamide) will be administered per os bi-daily (50 mg x 2), and given on a week on/ week off schedule.
  MK3475 will be administered intravenously (200 mg), and given every 3 weeks on day 8.
  G100 will be administered by intra-tumoral injection (20µg), one weekly injection for at least 6 weeks and for a maximum of 12 weeks. G100 will start one week before CP administration (impregnation phase).
  A treatment cycle consists of 3 weeks. Treatment may continue until disease progression or study discontinuation.
  Other Names: Pembrolizumab, Endoxan, GLA-SE (glucopyranosyl lipid adjuvant-stable emulsion).
  Arms: Stratum 7: Metastatic soft-tissue sarcoma.

SUMMARY:
This is a multicenter study assessing the efficacy of different therapeutic strategy in patients with advanced sarcomas.

DETAILED DESCRIPTION:
This is a phase 2 trial with 7 strata :

* Leiomyosarcoma (strata 1) : 33 patients
* Undifferentiated sarcoma (strata 2): 33 patients
* Sarcomas others (strata 3) : 33 patients
* Osteosarcoma (strata 4) : 33 patients
* GIST (strata 5): 31 patients
* Advanced soft-tissue sarcoma with immune signature (strata 6): 32 patients
* Metastatic soft-tissue sarcoma (strata 7): 32 patients

ELIGIBILITY:
Inclusion Criteria:

1. Histology : Leiomyosarcoma, or UPS, or other sarcoma, or GIST or osteosarcoma, or soft-tissue sarcoma with presence of tertiary lymphoid structures (stratum 6) histologically confirmed by central review.
2. Advanced non resectable / metastatic disease for strata 1 to 6. For stratum 7: locally advanced or metastatic disease with at least one injectable lesion.
3. Documented progression according to RECIST criteria. Progression on the last line of treatment should be confirmed by central review with two radiological assessments identical obtained at less than 6 months interval within the 12 months before inclusion.
4. For stratum 5, documented disease progression according to RECIST criteria after the first line imatinib and second line sunitinib.
5. Have provided tissue of a tumor lesion from an archival tissue sample obtained on metastasis or on locally advanced disease, or newly obtained core or excisional biopsy. For strata 6 and 7, tissue < 3 months old and with no subsequent treatment since or from a newly obtained biopsy.
6. For strata 1, 2, 3 and 6: no more of four previous lines of systemic therapy for metastatic disease and no more than 2 previous line for stratum 7.
7. Age ≥ 18 years.
8. ECOG performance status ≤ 1.
9. Measurable disease according to RECIST v1.1 outside any previously irradiated field. At least one site of disease must be uni-dimensionally ≥ 10 mm.
10. Life expectancy > 3 months (except for stratum 7 > 6 months).
11. ≥ 1 previous line (s) of chemotherapy in the palliative setting for strata 1 to 5. For other strata, participant must have advanced disease and must not be a candidate for other approved therapeutic regimen known to provide significant clinical benefit based on investigator judgement.
12. No symptomatic central nervous system disease.
13. No chronic use of glucocorticoids.
14. Adequate hematological, renal, metabolic and hepatic function:

    1. Hemoglobin ≥ 9 g/dl (patients may have received prior red blood cell transfusion); ANC ≥ 1.5 x 109/l and platelet count ≥ 100 x 109/l. For stratum 7: lymphocyte count ≥ 0.5.109 /l
    2. ALT and AST ≤ 2.5 x upper limit of normality (ULN) (≤ 5 in case of liver metastasis)
    3. Total bilirubin ≤ 1.5 x ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels ≥ 1.5 x ULN
    4. Albumin ≥ 25g/l
    5. Serum creatinine ≤ 1.5 x ULN OR CrCl ≥ 60 ml/min for subject with creatinine levels ≥ 1.5 x ULN,
    6. Creatine phosphokinase ≤ 2.5 x ULN
    7. INR ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
    8. aPTT ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
15. No prior or concurrent malignant disease diagnosed or treated in the last 2 years except for adequately treated in situ carcinoma of the cervix, basal or squamous skin cell carcinoma, or in situ transitional bladder cell carcinoma.
16. At least three weeks since last chemotherapy, immunotherapy or any other pharmacological treatment and/or radiotherapy.
17. Recovery to grade ≤ 1 from any adverse event from previous treatment (excluding alopecia of any grade and non-painful peripheral neuropathy grade ≤ 2 (NCI-CTCAE, v 4.0).
18. Women of childbearing potential must have a negative serum pregnancy test within 72 hours prior to receiving the first dose of study medication. Both women and men must agree to use a medically acceptable method of contraception throughout the treatment period and for four months after discontinuation of treatment. Acceptable methods for contraception include intrauterine device, oral contraceptive, subdermal implant and double barrier. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for ≥ 1 year.
19. Voluntary signed and dated written informed consents prior to any specific study procedure.
20. Patients with a French social security in compliance with the Law relating to biomedical research (Article 1121-11 of French Public Health Code).

Exclusion Criteria:

1. Previous treatment with MK3475 or CP or G100.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
3. Evidence of progressive or symptomatic central nervous system (CNS) or leptomeningeal metastases.
4. Men or women of childbearing potential who are not using an effective method of contraception as previously described; women who are pregnant or breast feeding.
5. Participation to a study involving a medical or therapeutic intervention in the last 30 days.
6. Previous enrolment in the present study.
7. Patient unable to follow and comply with the study procedures because of any geographical, familial, social or psychological reasons.
8. Known hypersensitivity to any involved study drug or of its formulation components.
9. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
10. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
11. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia, or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
12. Has known active hepatitis B or hepatitis C.
13. Has a known history of HIV (HIV1/2 antibodies).
14. Has received a live vaccine within 30 days prior to the first dose of trial treatment.
15. For strata 6 to 7:

    * patients with oral anticoagulation therapy
    * known urinary tract obstruction
    * previous allogenic bone marrow transplant
    * has an active infection requiring systemic treatment within 14 days prior to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2023-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine ITALIANO, MD, PhD, Study Chair — Institut Bergonié
Locations (8):
- France (8):
  - Institut Bergonié, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut Curie, Paris
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Toulmonde M, Penel N, Adam J, Chevreau C, Blay JY, Le Cesne A, Bompas E, Piperno-Neumann S, Cousin S, Grellety T, Ryckewaert T, Bessede A, Ghiringhelli F, Pulido M, Italiano A. Use of PD-1 Targeting, Macrophage Infiltration, and IDO Pathway Activation in Sarcomas: A Phase 2 Clinical Trial. JAMA Oncol. 2018 Jan 1;4(1):93-97. doi: 10.1001/jamaoncol.2017.1617. PMID 28662235
- [Result] Italiano A, Bessede A, Pulido M, Bompas E, Piperno-Neumann S, Chevreau C, Penel N, Bertucci F, Toulmonde M, Bellera C, Guegan JP, Rey C, Sautes-Fridman C, Bougouin A, Cantarel C, Kind M, Spalato M, Dadone-Montaudie B, Le Loarer F, Blay JY, Fridman WH. Pembrolizumab in soft-tissue sarcomas with tertiary lymphoid structures: a phase 2 PEMBROSARC trial cohort. Nat Med. 2022 Jun;28(6):1199-1206. doi: 10.1038/s41591-022-01821-3. Epub 2022 May 26. PMID 35618839
- [Result] Spalato-Ceruso M, Bouteiller F, Guegan JP, Toulmonde M, Bessede A, Kind M, Cousin S, Buy X, Palussiere J, Le Loarer F, Dadone-Montaudie B, Pulido M, Italiano A. Pembrolizumab combined with low-dose cyclophosphamide and intra-tumoral injection of the toll-like receptor 4 agonist G100 in patients with advanced pretreated soft tissue sarcoma: results from the PEMBROSARC basket study. J Hematol Oncol. 2022 Oct 27;15(1):157. doi: 10.1186/s13045-022-01377-2. PMID 36303228
- [Derived] Sun CM, Toulmonde M, Spalato-Ceruso M, Peyraud F, Bessede A, Kind M, Cousin S, Buy X, Palussiere J, Bougouin A, Sautes-Fridman C, Fridman HW, Pulido M, Italiano A. Impact of metronomic trabectedin combined with low-dose cyclophosphamide on sarcoma microenvironment and correlation with clinical outcome: results from the TARMIC study. Mol Cancer. 2024 Feb 19;23(1):37. doi: 10.1186/s12943-024-01942-y. PMID 38374062
- [Derived] Le Cesne A, Marec-Berard P, Blay JY, Gaspar N, Bertucci F, Penel N, Bompas E, Cousin S, Toulmonde M, Bessede A, Fridman WH, Sautes-Fridman C, Kind M, Le Loarer F, Pulido M, Italiano A. Programmed cell death 1 (PD-1) targeting in patients with advanced osteosarcomas: results from the PEMBROSARC study. Eur J Cancer. 2019 Sep;119:151-157. doi: 10.1016/j.ejca.2019.07.018. Epub 2019 Aug 21. PMID 31442817
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 8 centers:
  * Institut Bergonié, Pr Italiano
  * Centre Léon Bérard, Pr Blay
  * Institut Gustave Roussy, Dr Le Cesne
  * Centre Oscar Lambret, Dr Penel
  * Institut Curie, Dr Piperno-Neumann
  * Institut Paoli Calmette, Pr Bertucci
  * Institut Claudius Regaud, Dr Chevreau
  * Institut de Cancérologie de l'Ouest - Site René Gauducheau, Dr Bompas
  Planned enrollment period : 72 months Treatment duration : 2-years maximum Follow-up : 12 months Duration of study : 7 years
Groups:
- Stratum 1: Advanced Leiomyosarcoma; Stratum 2: Advanced Undifferentiated Sarcoma; Stratum 3: Advanced Other Sarcoma; Stratum 4: Advanced GIST; Stratum 5: Advanced Soft-tissue Sarcomas; Stratum 6: Advanced Soft-tissue Sarcomas With Immune Signature: Treatment strategy A: Combination of MK3475 with Metronomic CP administered to patients with advanced leiomyosarcoma.
  MK3475 will be administered intraveinously. Metronomic CP (Cyclophosphamide) will be adminstered orally.
  Combination of MK3475 with Metronomic CP:
  Metronomic CP (cyclophosphamide) will be administered per os bi-daily (50 mg x 2), and given on a week on/ week off schedule.
  MK3475 will be administered intraveinously (200mg in 30 minutes -5 min/+10 min) and given every 3 weeks on day 8.
  A treatment cycle consists of 3 weeks. Treatment may continue until disease progression or study discontinuation.
- Stratum 7: Metastatic Soft-tissue Sarcoma.: Treatment strategy B: Combination of MK3475 with Metronomic CP and G100. MK3475 will be administered intravenously. Metronomic CP (Cyclophosphamide) will be administered orally. G100 will be administered by intra-tumoral injection.
  Combination of MK3475 with Metronomic CP and G100:
  Metronomic CP (cyclophosphamide) will be administered per os bi-daily (50 mg x 2), and given on a week on/ week off schedule.
  MK3475 will be administered intraveinously (200mg in 30 minutes -5 min/+10 min) and given every 3 weeks on day 8.
  G100 will be administered by intra-tumoral injection (20µg), one weekly injection for at least 6 weeks and for a maximum of 12 weeks. G100 will start one week before CP administration (impregnation phase).
  A treatment cycle consists of 3 weeks. Treatment may continue until disease progression or study discontinuation.
Period: Overall Study
Arm/Group | Stratum 1: Advanced Leiomyosarcoma | Stratum 2: Advanced Undifferentiated Sarcoma | Stratum 3: Advanced Other Sarcoma | Stratum 4: Advanced GIST | Stratum 5: Advanced Soft-tissue Sarcomas | Stratum 6: Advanced Soft-tissue Sarcomas With Immune Signature | Stratum 7: Metastatic Soft-tissue Sarcoma.
Started | 15 | 16 | 16 | 17 | 10 | 35 | 20
Completed | 13 | 14 | 14 | 15 | 9 | 30 | 17
Not Completed | 2 | 2 | 2 | 2 | 1 | 5 | 3
Not completed — Protocol Violation | 2 | 2 | 2 | 2 | 1 | 5 | 3

BASELINE CHARACTERISTICS:
Population: * Eligible population: All patients included without major violation of eligibility criteria.
  * Population eligible and assessable for the primary endpoint : eligible patients who received at least one administration of PEMBROLIZUMAB and one administration of Metronomic CP
  * Safety population: All patients with at least one treatment (any) administration.
Groups:
- Stratum 7: Metastatic Soft-tissue Sarcoma.: Treatment strategy B: Combination of MK3475 with Metronomic CP and G100. MK3475 will be administered intravenously . Metronomic CP (Cyclophosphamide) will be administered orally. G100 will be administered by intra-tumoral injection.
  Combination of MK3475 with Metronomic CP and G100:
  Metronomic CP (cyclophosphamide) will be administered per os bi-daily (50 mg x 2), and given on a week on/ week off schedule.
  MK3475 will be administered intraveinously (200mg in 30 minutes -5 min/+10 min) and given every 3 weeks on day 8.
  G100 will be administered by intra-tumoral injection (20µg), one weekly injection for at least 6 weeks and for a maximum of 12 weeks. G100 will start one week before CP administration (impregnation phase).
  A treatment cycle consists of 3 weeks. Treatment may continue until disease progression or study discontinuation.
- Total: Total of all reporting groups
Arm/Group | Stratum 1: Advanced Leiomyosarcoma | Stratum 2: Advanced Undifferentiated Sarcoma | Stratum 3: Advanced Other Sarcoma | Stratum 4: Advanced GIST | Stratum 5: Advanced Soft-tissue Sarcomas | Stratum 6: Advanced Soft-tissue Sarcomas With Immune Signature | Stratum 7: Metastatic Soft-tissue Sarcoma. | Total
Number analyzed (Participants) | 15 | 16 | 16 | 17 | 10 | 35 | 20 | 129
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 63.7 [56.8 to 72.2] | 59.1 [55.9 to 64.4] | 55.5 [45.4 to 60.1] | 42.2 [22.3 to 52.0] | 57.9 [44.3 to 69.9] | 62.2 [45.2 to 77.1] | 62.7 [57.0 to 69.0] | 63 [57 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 6 | 7 | 5 | 16 | 10 | 57
  Male | 7 | 11 | 10 | 10 | 5 | 19 | 10 | 72
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 15 | 16 | 16 | 17 | 10 | 35 | 20 | 129

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Objective Response at 6 Months
Description: Objective response is defined according to RECIST v1.1 as either complete response (disappearance of all target lesions, with any pathological lymph nodes reduced in short axis to <10 mm) or partial response (≥30% decrease in the sum of diameters of target lesions compared with baseline).
  This primary endpoint is part of a dual endpoint encompassing both non-progression and objective response at 6 months (non-progression is presented as a separate primary outcome). ORR at 6 months will be evaluated only in the following strata: Stratum 1: Advanced leiomyosarcoma ; Stratum 2: Advanced undifferentiated sarcoma ; Stratum 3: Advanced other sarcoma ; Stratum 4: Advanced osteosarcoma
Time Frame: 6 months from treatment initiation
Population: Population eligible and assessable for the primary endpoint: eligible patients who received at least one administration of PEMBROLIZUMAB and one administration of Metronomic CP.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Stratum 4: Advanced Osteosarcoma: Treatment strategy A: Combination of MK3475 with Metronomic CP administered to patients with advanced leiomyosarcoma.
  MK3475 will be administered intraveinously. Metronomic CP (Cyclophosphamide) will be adminstered orally.
  Combination of MK3475 with Metronomic CP:
  Metronomic CP (cyclophosphamide) will be administered per os bi-daily (50 mg x 2), and given on a week on/ week off schedule.
  MK3475 will be administered intraveinously (200mg in 30 minutes -5 min/+10 min) and given every 3 weeks on day 8.
  A treatment cycle consists of 3 weeks. Treatment may continue until disease progression or study discontinuation.
Arm/Group | Stratum 1: Advanced Leiomyosarcoma | Stratum 2: Advanced Undifferentiated Sarcoma | Stratum 3: Advanced Other Sarcoma | Stratum 4: Advanced Osteosarcoma
Number analyzed (Participants) | 13 | 14 | 14 | 15
percentage of participants | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 6.7 [0.2 to 32.0]

2. Primary Outcome: Percentage of Particpants in Non-progression at 6 Months
Description: Non-progression is defined as the absence of progressive disease according to RECIST v1.1. Progressive disease defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
  This outcome will be assessed as a stand-alone primary endpoint in the following strata: Stratum 5: Advanced gastrointestinal stromal tumor (GIST) ; Stratum 6: Advanced soft tissue sarcomas with immune signature ; Stratum 7: Metastatic soft tissue sarcoma (STS)
  In strata 1 to 4, non-progression is considered as part of the dual primary endpoint together with objective response at 6 months.
Time Frame: 6 months from treatment initiation
Population: Population eligible and assessable for the primary endpoint: eligible patients who received at least:
  * For all strata (except for stratum 7): one administration of PEMBROLIZUMAB and one administration of Metronomic CP
  * For stratum 7: one administration of PEMBROLIZUMAB and one administration of Metronomic CP and one administration of G100.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stratum 1: Advanced Leiomyosarcoma | Stratum 2: Advanced Undifferentiated Sarcoma | Stratum 3: Advanced Other Sarcoma | Stratum 4: Advanced GIST | Stratum 5: Advanced Soft-tissue Sarcomas | Stratum 6: Advanced Soft-tissue Sarcomas With Immune Signature | Stratum 7: Metastatic Soft-tissue Sarcoma.
Number analyzed (Participants) | 13 | 14 | 14 | 15 | 9 | 30 | 17
percentage of participants | 0.0 [0.0 to 0.0] | 7.1 [0.2 to 33.9] | 14.3 [1.8 to 42.8] | 13.3 [1.7 to 40.5] | 11.1 [2.8 to 48.3] | 40 [22.7 to 59.4] | 11.8 [1.5 to 36.4]

3. Secondary Outcome: Percentage of Patients Remaining Alive With Best Overall Response as Per RECIST v1.1.
Description: Best overall response is defined as the best response across all time points (RECIST v1.1). The best overall response is determined once all the data for the participant is known.
  Each patient has been assigned one of the following categories (RECIST 1.1): complete response (disappearance of all target lesions); partial response (>=30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters); progression (20% increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) and stable disease (nor CR, PR or progression).
Time Frame: 6 months from treatment initiation
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stratum 1: Advanced Leiomyosarcoma | Stratum 2: Advanced Undifferentiated Sarcoma | Stratum 3: Advanced Other Sarcoma | Stratum 4: Advanced GIST | Stratum 5: Advanced Soft-tissue Sarcomas | Stratum 6: Advanced Soft-tissue Sarcomas With Immune Signature | Stratum 7: Metastatic Soft-tissue Sarcoma.
Number analyzed (Participants) | 13 | 14 | 14 | 15 | 9 | 30 | 17
percentage of participants
  Complete response (CR) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Partial response (PR) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 6.7 [0.2 to 32.0] | 0 [0 to 0] | 26.7 [12.3 to 45.9] | 5.9 [0.2 to 28.7]
  Stable disease (SD) | 23.1 [5.0 to 53.8] | 35.7 [12.8 to 64.9] | 35.7 [12.8 to 64.9] | 33.3 [11.8 to 61.6] | 33.3 [7.5 to 70.1] | 36.7 [19.9 to 56.1] | 23.5 [6.8 to 49.9]
  Progression (PD) | 76.9 [46.2 to 95.0] | 50.0 [23.0 to 77.0] | 57.1 [28.9 to 82.3] | 53.3 [26.6 to 78.7] | 66.7 [29.9 to 92.5] | 33.3 [17.3 to 52.8] | 70.6 [44.0 to 89.7]
  Not evaluable for response (NE) | 0 [0 to 0] | 14.3 [1.8 to 42.8] | 7.1 [0.2 to 33.9] | 6.7 [0.2 to 32.0] | 0 [0 to 0] | 3.3 [0.1 to 17.2] | 0 [0 to 0]

4. Secondary Outcome: Median Progression-free Survival
Description: Progression-free survival (PFS) is defined as the time from study treatment initiation to the first occurrence of disease progression or death (of any cause), whichever occurs first.
  Progressive disease defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
  Patients alive and progression free were censored at the date of last follow-up, death, or last patient contact. Progression is assessed as per RECIST v1.1.
  Progression-free survival is estimated as a function of time using Kaplan-Meier method.
Time Frame: From start of treatment, and during treatment until progression or death for any cause, whichever occurs first, for up to 12 months.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stratum 1: Advanced Leiomyosarcoma | Stratum 2: Advanced Undifferentiated Sarcoma | Stratum 3: Advanced Other Sarcoma | Stratum 4: Advanced GIST | Stratum 5: Advanced Soft-tissue Sarcomas | Stratum 6: Advanced Soft-tissue Sarcomas With Immune Signature | Stratum 7: Metastatic Soft-tissue Sarcoma.
Number analyzed (Participants) | 13 | 14 | 14 | 15 | 9 | 30 | 17
months | 1.4 [1.2 to 1.4] | 1.3 [1.1 to 2.9] | 1.4 [0.9 to 4.0] | 1.4 [1.0 to 1.4] | 1.4 [0.9 to 5.3] | 4.1 [1.4 to 12.5] | 1.8 [1.5 to 4.1]

5. Secondary Outcome: Median Overall Survival
Description: Overall survival (OS) defined as the time from randomization to death (due to any cause). Patients alive were censored at the date of last follow-up or last patient contact. Overall survival was estimated as a function of time using Kaplan-Meier method.
Time Frame: From start of treatment, and during treatment until death for any cause for up to 30 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stratum 1: Advanced Leiomyosarcoma | Stratum 2: Advanced Undifferentiated Sarcoma | Stratum 3: Advanced Other Sarcoma | Stratum 4: Advanced GIST | Stratum 5: Advanced Soft-tissue Sarcomas | Stratum 6: Advanced Soft-tissue Sarcomas With Immune Signature | Stratum 7: Metastatic Soft-tissue Sarcoma.
Number analyzed (Participants) | 13 | 14 | 14 | 15 | 9 | 30 | 17
months | 15.1 [4.4 to 17.9] | 6.7 [3.2 to 20.0] | 7.1 [2.0 to 16.3] | 5.6 [2.1 to 12.1] | NA [NA to NA] — The median overall survival was not reached, as fewer than 50% of patients had experienced the event at the time of analysis. | 18.3 [8.5 to NA] — The median overall survival was estimated at 18.3 months (95% CI: 8.5 - NA). The upper bound of the confidence interval could not be determined due to an insufficient number of deaths occurring after the median time | 25.2 [8.5 to NA] — The median overall survival was 25.2 months. The upper bound of the confidence interval could not be estimated (noted as "NR" for "Not Reached") due to the limited number of events after the median and the small sample size.

ADVERSE EVENTS:
Time Frame: Adverse events (serious and non-serious) and deaths were reported for 90 days after the last treatment administration or until the start of a new antitumor therapy, whichever occurs first, up to 30 months.
Description: Safety population: All patients with at least one treatment (any) administration.
Groups:
- Stratum 1: Advanced Leiomyosarcoma: Treatment strategy A:
  Combination of MK3475 with Metronomic CP administered to patients with advanced leiomyosarcoma.
  MK3475 will be administered intraveinously. Metronomic CP (Cyclophosphamide) will be adminstered orally.
  Combination of MK3475 with Metronomic CP:
  Metronomic CP (cyclophosphamide) will be administered per os bi-daily (50 mg x 2), and given on a week on/ week off schedule.
  MK3475 will be administered intraveinously, and given every 3 weeks on day 8. A treatment cycle consists of 3 weeks. Treatment may continue until disease progression or study discontinuation.
- Stratum 2: Advanced Undifferentiated Sarcoma: Treatment strategy A:
  Combination of MK3475 with Metronomic CP administered to patients with advanced undifferentiated sarcoma.
  MK3475 will be administered intraveinously. Metronomic CP (Cyclophosphamide) will be adminstered orally.
  Combination of MK3475 with Metronomic CP:
  Metronomic CP (cyclophosphamide) will be administered per os bi-daily (50 mg x 2), and given on a week on/ week off schedule.
  MK3475 will be administered intraveinously, and given every 3 weeks on day 8. A treatment cycle consists of 3 weeks. Treatment may continue until disease progression or study discontinuation.
- Stratum 3: Advanced Other Sarcoma: Treatment strategy A:
  Combination of MK3475 with Metronomic CP administered to patients with advanced other sarcoma.
  MK3475 will be administered intraveinously. Metronomic CP (Cyclophosphamide) will be adminstered orally.
  Combination of MK3475 with Metronomic CP:
  Metronomic CP (cyclophosphamide) will be administered per os bi-daily (50 mg x 2), and given on a week on/ week off schedule.
  MK3475 will be administered intraveinously, and given every 3 weeks on day 8. A treatment cycle consists of 3 weeks. Treatment may continue until disease progression or study discontinuation.
- Stratum 4: Advanced GIST: Treatment strategy A:
  Combination of MK3475 with Metronomic CP administered to patients with advanced GIST.
  MK3475 will be administered intraveinously. Metronomic CP (Cyclophosphamide) will be adminstered orally.
  Combination of MK3475 with Metronomic CP:
  Metronomic CP (cyclophosphamide) will be administered per os bi-daily (50 mg x 2), and given on a week on/ week off schedule.
  MK3475 will be administered intraveinously, and given every 3 weeks on day 8. A treatment cycle consists of 3 weeks. Treatment may continue until disease progression or study discontinuation.
- Stratum 5: Advanced Soft-tissue Sarcomas: Treatment strategy A:
  Combination of MK3475 with Metronomic CP administered to patients with advanced soft-tissue sarcomas.
  MK3475 will be administered intraveinously. Metronomic CP (Cyclophosphamide) will be adminstered orally.
  Combination of MK3475 with Metronomic CP:
  Metronomic CP (cyclophosphamide) will be administered per os bi-daily (50 mg x 2), and given on a week on/ week off schedule.
  MK3475 will be administered intraveinously, and given every 3 weeks on day 8. A treatment cycle consists of 3 weeks. Treatment may continue until disease progression or study discontinuation.
- Stratum 6: Advanced Soft-tissue Sarcomas With Immune Signature: Treatment strategy A:
  Combination of MK3475 with Metronomic CP administered to patients with advanced soft-tissue sarcomas with immune signature.
  MK3475 will be administered intraveinously. Metronomic CP (Cyclophosphamide) will be adminstered orally.
  Combination of MK3475 with Metronomic CP:
  Metronomic CP (cyclophosphamide) will be administered per os bi-daily (50 mg x 2), and given on a week on/ week off schedule.
  MK3475 will be administered intraveinously, and given every 3 weeks on day 8. A treatment cycle consists of 3 weeks. Treatment may continue until disease progression or study discontinuation.
- Stratum 7: Metastatic Soft-tissue Sarcoma.: Treatment strategy B:
  Combination of MK3475 with Metronomic CP and G100. MK3475 will be administered intravenously. Metronomic CP (Cyclophosphamide) will be administered orally. G100 will be administered by intra-tumoral injection.
  Combination of MK3475 with Metronomic CP:
  Metronomic CP (cyclophosphamide) will be administered per os bi-daily (50 mg x 2), and given on a week on/ week off schedule.
  MK3475 will be administered intraveinously, and given every 3 weeks on day 8. A treatment cycle consists of 3 weeks. Treatment may continue until disease progression or study discontinuation.
Arm/Group | Stratum 1: Advanced Leiomyosarcoma | Stratum 2: Advanced Undifferentiated Sarcoma | Stratum 3: Advanced Other Sarcoma | Stratum 4: Advanced GIST | Stratum 5: Advanced Soft-tissue Sarcomas | Stratum 6: Advanced Soft-tissue Sarcomas With Immune Signature | Stratum 7: Metastatic Soft-tissue Sarcoma.
All-Cause Mortality (participants affected / at risk) | 13/15 | 14/16 | 7/16 | 12/16 | 3/10 | 15/35 | 9/19
Serious Adverse Events (participants affected / at risk) | 5/15 | 10/16 | 9/16 | 12/16 | 9/10 | 14/35 | 8/19
Other Adverse Events (participants affected / at risk) | 15/15 | 16/16 | 16/16 | 16/16 | 10/10 | 35/35 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1: Advanced Leiomyosarcoma (N=15) | Stratum 2: Advanced Undifferentiated Sarcoma (N=16) | Stratum 3: Advanced Other Sarcoma (N=16) | Stratum 4: Advanced GIST (N=16) | Stratum 5: Advanced Soft-tissue Sarcomas (N=10) | Stratum 6: Advanced Soft-tissue Sarcomas With Immune Signature (N=35) | Stratum 7: Metastatic Soft-tissue Sarcoma. (N=19)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 1 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
General disorders and administration site conditions (General disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic hemorrhage (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Spesis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocytes count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other, specif (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (4) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Edema cerebral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1: Advanced Leiomyosarcoma (N=15) | Stratum 2: Advanced Undifferentiated Sarcoma (N=16) | Stratum 3: Advanced Other Sarcoma (N=16) | Stratum 4: Advanced GIST (N=16) | Stratum 5: Advanced Soft-tissue Sarcomas (N=10) | Stratum 6: Advanced Soft-tissue Sarcomas With Immune Signature (N=35) | Stratum 7: Metastatic Soft-tissue Sarcoma. (N=19)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4) | 9 (11) | 4 (4) | 2 (4) | 8 (8) | 5 (5)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 8 (8) | 1 (1)
Conjonctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 7 (8) | 3 (3)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 6 (6) | 3 (3)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 5 (9) | 1 (1) | 1 (1) | 10 (11) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3) | 4 (6) | 2 (3) | 13 (13) | 9 (9)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 3 (3) | 4 (4)
Chill (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (5) | 2 (2) | 4 (4) | 2 (2)
Fatigue (General disorders) | 11 (12) | 7 (7) | 11 (13) | 8 (9) | 9 (10) | 23 (24) | 10 (10)
Fever (General disorders) | 1 (1) | 2 (2) | 2 (3) | 1 (1) | 3 (5) | 4 (4) | 1 (1)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (2) | 1 (1) | 0 (0) | 6 (7) | 2 (2) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other, specifiy (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Autoimmune disorder (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 2 (5) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Lip infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Rhinitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (5) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 6 (8) | 3 (3)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 4 (4) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CPK increase (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
GGT increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 3 (3) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 16 (16) | 7 (7)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 2 (2)
Weight loss (Investigations) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 6 (6) | 4 (4) | 4 (4) | 3 (3) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 1 (1) | 2 (4) | 1 (1) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (4) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 3 (3) | 2 (3) | 0 (0) | 6 (7) | 10 (12)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Ohter, specify (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Phantom pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 2 (2) | 2 (2) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (5) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 5 (6) | 4 (4) | 1 (2) | 3 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (5) | 1 (2) | 1 (1) | 2 (2)
Sinus disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hyperrhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 4 (5) | 3 (3) | 0 (0) | 4 (6) | 2 (2)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT02406781/Prot_000.pdf
  • Statistical Analysis Plan (2015-12-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT02406781/SAP_001.pdf